CLINICAL TRIAL: NCT00750022
Title: Feasibility Study of Integrating IC Technology With the WatchWT Comprehensive Weight Reduction Program.
Brief Title: Feasibility of Integrating Indirect Calorimetry (IC) Technology in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado Center for Chronic Care Innovations, Inc. (Other)
Collaborators: Microlife Medical Home Solutions, Inc. (Industry)
Responsible Party: Scott McDoniel; Director of Clinical Affairs, Microlife Medical Home Solutions, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WCPC-0101
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Obesity; Hypertension
MeSH Terms: conditions — Obesity; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- E1 (Experimental)
  Interventions: Behavioral: Usual Care
- A1 (Active Comparator)
  Interventions: Behavioral: Individualized IC treatment

INTERVENTIONS:
Behavioral: Individualized IC treatment — Individuals will receive IC measurement at baseline and three months. Nutrition and physical activity plan will be developed and adjusted from measured RMR and lifestyle.
  Other Names: MedGem indirect Calorimeter
  Arms: A1
Behavioral: Usual Care — Individuals will receive standard dietary plan. Women will receive 1200 Kcal/day and men will receive 1600 Kcal/day. Individuals will receive RMR measurement at three months. RMR information will be used to help improve eating behavior.
  Other Names: MedGem indirect Calorimeter
  Arms: E1

SUMMARY:
The purpose of this study is to evaluate the feasibility of using indirect calorimetry (IC) within a comprehensive weight reduction program. Will individuals that receive a personalized nutrition program, at baseline, from IC technology respond better to treatment compared to individuals receiving IC technology at three months.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than 30 kg/m2
* 18-70 years of age

Exclusion Criteria:

* No participation in other weight loss efforts outside study.
* Pregnant or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Bodyweight | Six Months

SECONDARY OUTCOMES:
Psychobehavioral: Self-Efficacy | Six Months
Quality Life | Six Months
Blood Pressure | Six Months
Eating Behavior | Six Months

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado Center for Chronic Care Innovations, Westminster, Colorado, United States

REFERENCES:
- [Derived] McDoniel SO, Wolskee P, Shen J. Treating obesity with a novel hand-held device, computer software program, and Internet technology in primary care: the SMART motivational trial. Patient Educ Couns. 2010 May;79(2):185-91. doi: 10.1016/j.pec.2009.07.034. Epub 2009 Aug 20. PMID 19699049